CLINICAL TRIAL: NCT05084157
Title: Prospective, Multicentre, International, Registry of LONG-term Findings at Cardiac Imaging in TAKotsubo SyndromE (The LONG-TAKE Registry)
Brief Title: Long-term Echocardiographic Findings in Takotsubo Syndrome
Acronym: LONG-TAKE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Associate Professor, University of Roma La Sapienza
Other Study IDs: D-21-1111
Record Dates: First submitted 2021-10-05; First posted 2021-10-19 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Takotsubo Cardiomyopathy
Keywords: syndrome
MeSH Terms: conditions — Takotsubo Cardiomyopathy; Syndrome | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Echocardiography — Patients will undergo Doppler echocardiography

SUMMARY:
Takotsubo syndrome (TTS) is characterized by severe left ventricular (LV) dysfunction that gradually recovers, thus leading to the commonly accepted belief that it is a transient and self-limiting condition.

Histologically, TTS can be accompanied by severe morphological alterations potentially resulting from catecholamine excess followed by microcirculatory dysfunction and direct cardiotoxicity. The affected myocardium, however, has a high potential of structural reconstitution which correlates with the rapid functional recovery. The lack of persistent morphological changes in TTS has been confirmed by original CMR studies which pointed out that the acute phase of the disease is characterized only by remarkable myocardial edema with no evidence of significant late gadolinium enhancement. Indeed, the absence of LGE in TTS patients has become a common diagnostic criterion in most CMR centers. Although some studies have challenged this notion by reporting delayed hyper-enhancement in TTS patients, the intensity and extent of LGE in the acute phase of TTS are less than usually reported in studies of myocardial infarction.

The long-term clinical and functional consequences of an acute episode of TTS are still unclear. A recent spectroscopic investigation has shown that long-term (>1 year) abnormalities in cardiac energetic persist after an acute episode of TTS. Also, a few patients with residual wall motion abnormality in whom LGE fails to resolve (suggesting the acute event resulted in frank infarction) have been reported. However, how often persistent morphologic abnormalities are present after the index episode remains undefined. The possibility exists that fibrosis was undetected at follow-up CMR studies using conventional LGE threshold methods due to the fact that myocardial injury is subtler and there are no confidently recognizable reference regions of normal myocardium. Newer echocardiographic tools (i.e. tissue Doppler) have now the potential to detect persistence of post-TTS LV function abnormalities.

DETAILED DESCRIPTION:
Objective of the study The aim of this study is to assess the frequency of long-term (>12 months) morphologic abnormalities at cardiac imaging after an index episode of TTS, and their possible correlation with presenting features and long-term outcome

Study Population The registry will enrol consecutive patients with TS who have undergone echocardiography either at entry and during follow-up (>12 months).

Registry Design This is a non-interventional, multi-centre, registry of male and female patients with TTS who undergo follow-up echocardiography after the index event.

Rationale This large global registry focuses on long-term findings in TTS patients. The registry is observational, and decisions on patient management are determined by the health care professional and the patient and not by the protocol. Patients are therefore treated according to normal local practice.

Source Data: Data will be derived from the patients clinical records according to specifications outlined in the electronic case report form. This Registry will not undertake any experimental intervention with patients being treated according to normal local practice. No additional tests or procedures are required by the protocol. Physicians involved in initial diagnosis of TTS in patients may transfer or refer the cases to other physicians who will treat and follow up the patients in the long-term.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of TTS according to current International consensus criteria
* Written informed consent
* Age 18 years and over

Exclusion Criteria:

* Secondary form of TTS (e.g. as it can occur after sepsis, neurological disorders, pheochromocytoma)
* Durg-induced form of TTS (e.g. after administration of drugs such as dopamine, dobutamine, epinephrine, or norepinephrine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as having Takotsubo Syndrome on the basis of Mayo Criteria
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Left ventricular systolic dysfunction | Up to 5 years
  The time to the echocardiographic finding of left ventricular systolic dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Gaudio, MD, Study Chair — University Sapienza

IPD SHARING:
Plan to Share IPD: Undecided